CLINICAL TRIAL: NCT05595837
Title: Immune Registry for Organ Transplantation From COVID Positive Donors.
Status: Completed | Type: Observational
Sponsor: Virginia Commonwealth University (Other)
Collaborators: Eurofins (Industry)
Responsible Party: Sponsor
Other Study IDs: HM20024454
Record Dates: First submitted 2022-10-20; First posted 2022-10-27 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: COVID-19; Organ Transplant
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COVID-19 positive donors
  Interventions: Other: Standard organ transplant
- COVID-19 negative donors
  Interventions: Other: Standard organ transplant

INTERVENTIONS:
Other: Standard organ transplant — Standard organ transplant procedures and follow up care

SUMMARY:
The purpose of this study is to collect data generated by standard clinical practice to determine the short term and long term clinical outcomes of recipients of solid organ transplantation from COVID-19 infected donors and compare it to recipients with organ transplant from COVID-19 negative donors.

DETAILED DESCRIPTION:
To advance science, it is helpful for researchers to share information. They do this by putting data or biospecimens into one or more scientific databases (called registries or repositories), where it is stored along with information from other studies. Researchers can then study the information in other ways and combine information from many studies to learn even more. The researchers are asking for permission to store and share personal information in a research registry to help research studies in the future. The information will be available for any research question, such as research to understand what causes certain diseases in patients with solid organ transplant, development of new scientific methods, or the study of where different groups of people may have come from.

Information from participant's medical chart will be securely stored in the VCU database. This will include donor information (including COVID test results, radiologic findings, symptoms, treatments, cause of death etc.) as well as recipient information (including demographics, labs, biopsy findings if any, length of hospital stay, COVID transmission, graft function, immunosuppression, post-transplant complications and long term clinical outcomes like patient and graft survival, etc.). Data will be collected during routine clinical care.

The study will include the following tests:

* Pre transplant COVID-19 PCR on the nasal swab (as standard transplant protocol), serum COVID-19 specific T-cell immune response, and serum COVID-19 spike antibody as a study protocol in all the recipients.
* Posttransplant COVID-19 spike antibody in the serum around 4 weeks after the completion of induction Thymoglobulin as a study protocol in all the recipients.
* Daily COVID-19 PCR in serum from post-operative day 1 till post-operative day 4 as a study protocol in the recipients with organ transplant from COVID-19 positive donors.
* Posttransplant COVID-19 PCR nasal swab once around one-week post-transplant as study protocol in the recipients with organ transplant from COVID-19 positive donors.
* COVID-19 T-cell specific immune response will be checked in the recipient's serum at 4 weeks post-transplant as study protocol in all the recipients.
* According to the standard transplant protocol post-transplant donor-specific antibodies will be checked around 2 weeks post transplant and the results will direct the donor-derived cell-free DNA testing in all the recipients.

ELIGIBILITY:
Inclusion Criteria:

- Adult (>18 years old) male and female solid organ transplant recipients

Exclusion Criteria:

* Absence of informed consent for the clinical protocol and the registry.
* Prisoners will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Solid organ transplant recipients
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2022-12-29 (Actual); Primary Completion 2025-07-20 (Actual); Study Completion 2025-07-20 (Actual)

PRIMARY OUTCOMES:
Number of participants who test positive for COVID-19 | 1 week post transplant
Serum COVID-19 T-cell specific immune response | 4 week post transplant
  Blood samples from participants will be tested for the presence or absence of COVID-19 immune response markers, i.e. T-cells. The existence of T-cells will be marked as positive, indicating an immune response in the participant to COVID-19.

CONTACTS AND LOCATIONS:
Overall Officials: Ambreen Azhar, MD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No